CLINICAL TRIAL: NCT04495348
Title: Explorations Into the Mechanism for INSTI-associated Weight Gain: a Focus on Energy Balance
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-2960
Record Dates: First submitted 2020-07-17; First posted 2020-07-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: HIV-1-infection; Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — doravirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open-label arm: Participants are switched to doravirine and then switched back to INSTI-based therapy.
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Participants will be switched to doravirine and then switched back to INSTI-based therapy to determine the impact on energy balance.

SUMMARY:
Weight gain following antiretroviral therapy (ART) initiation occurs with all modern regimens. Recent real-world reports suggest that integrase strand transfer inhibitor (INSTI)-based ART may be associated with excess weight gain compared to other regimens. Weight gain appears to occur regardless of baseline weight, and is most pronounced among women and minorities, often those at highest risk of obesity-associated comorbidities. INSTI- and TAF-based regimens are now preferred regimens for most persons according to the Department of Health and Human Services ART-Treatment Guidelines. As a result, there is an urgent need to understand the underlying mechanisms for this weight gain.

This study aims to understand the changes in energy balance that occur with changes in ART. Participants with HIV who have experienced >10% weight gain on INSTI (bictegravir or dolutegravir-based therapy) will be switched to doravirine for 12 weeks, and then back to their prior INSTI regimen, allowing for assessment of changes in metabolic parameters with drug withdrawal and reintroduction (with no change to NRTI-backbone). Twenty-four hour energy balance will be measured on both regimens during a 24-hour stay using a whole room indirect calorimetry, with a standardized diet. Ultimately, the investigator's goal is to understand the mechanisms of weight gain so that future interventions can most effectively mitigate ART-associated weight changes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >=18 years
* BMI of >=30.0 kg/m2
* >=10% weight gain within the first 2 years of switching to INSTI-based ART (bictegravir or dolutegravir-based regimens only), with weight gain that has continued or worsened (not decreased).
* At least one plasma HIV-1 RNA <50 copies/mL while on the current INSTI-based ART within 6 months of screening
* Willing to switch to doravirine and pay any associated co-pays that may not be covered by insurance.
* NRTI back-bone therapy with either TAF or TDF with 3TC or FTC and willing to continue these 2 agents

Exclusion Criteria:

* Use of an INSTI other than bictegravir or dolutegravir within the 1 year prior to entry
* Any plasma HIV-1 RNA >500 copies/mL within one year prior to entry
* Pregnant, breast-feeding, or intention to become pregnant during the study period.
* Participants using medications with a potential serious drug-drug interaction with doravirine that cannot be attenuated through dose change will also be excluded.
* Any plans to change diet or exercise regimen significantly within the study period.

NOTE: Significantly refers to intent to join a weight-loss program such as Weight Watchers, start a specific diet (such as ketogenic or very low carbohydrate).

- Use of human growth hormone, tesamorelin, supra-physiologic testosterone to achieve therapeutic blood levels, or any use of other anabolic steroids within 3 months prior to study entry or plans to start these on study.

NOTE: Chronic, stable hormone replacement therapy ≥3 months prior to entry in men with diagnosed hypogonadism or transgender person on masculinizing hormonal therapy is permitted.

- Use of estrogens or progesterones at supraphysiologic doses within 3 months prior to study entry.

NOTE: Stable doses used for contraception, post-menopausal hormone replacement or feminizing hormone therapy for transgender persons ≥3 months prior to entry is permitted.

* Use of prednisone (or equivalent steroid) within the prior 3 months, unless stable dosing ≤ 10mg
* Change or initiation of lipid- and/or glucose-lowering therapy in the 12 weeks prior to entry, or planned need for such therapy during the study period. Use of stable lipid- and/or glucose-lowering therapy during the study is allowed.
* Current serious illness requiring systemic treatment and/or hospitalization until participant completes therapy or is clinically stable as determined by the site investigator.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Intent to use any medication likely to cause significant changes in weight during the study period.

NOTE: A list of medications in this category will be provided.

* Prior bariatric surgery (e.g., lap band, gastric sleeve, or roux-en-y bypass surgery) or major gastric surgery or plans to undergo weight reduction surgery while on study.
* Screening laboratory values as follows:

ANC < 500 cells/mm3 Hemoglobin < 9 gm/dL Cr Cl < 30 mL/min (estimated by CKD-Epi equation) Fasting blood sugar <200

* Any chronic, end-stage organ disease that would impact metabolism, including end-stage liver or renal disease, cardiac cachexia, chronic obstructive pulmonary disease, or cancer
* Any condition that the study investigator believes would make the candidate unsuitable for participation.
* Severe claustrophobia that would limit ability of participant to remain in the whole room calorimeter
* Known resistance to any component of the study drugs, including detection of any of the following resistance mutations on prior HIV genotype test (genotype testing not required if not available): Doravirine resistance: V106A, V106I, V106T, V106M, Y188C, Y188H, Y188L, G190E, P225H, F227C, F227L, F227R, M230L, L234I Resistance to NRTIs: K65R, K65E, K65N, T69S (insertion complex), K70E, L74V, Y115F, Q151M, M184I, M184V.
* Active severe depression or anxiety, as evidenced by recent inpatient psychiatric admission (within the prior 6 months); PHQ-2 score of 6 (response of 'nearly every day' to 'do you have little interest or pleasure in doing things' or 'feeling down, depressed, or hopeless'; expressed suicidal ideations.
* Under the care of a provider for disordered eating (bulimia, anorexia, or other).
* Diabetes will be permitted if well-controlled with a Hb A1C of 7.5% of less in the prior 6 months and no use of insulin.
* Routine physical activity meeting or exceeding 150 minutes/week of moderate or vigorous activity, for at least 3 months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HIV who have experienced >10% weight gain on INSTI (bictegravir or dolutegravir-based therapy).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change in energy balance | 24 weeks
  Change in total energy expenditure (kcal/day)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Erlandson, MD, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UTHealth, Houston, Texas

IPD SHARING:
Plan to Share IPD: No